CLINICAL TRIAL: NCT03177434
Title: Multicenter Study Evaluating the Efficacy of Dicopeg Junior in Comparison With Lactulose for the Treatment of Functional Constipation in Children Aged 6 Months to 6 Years. A Prospective, Randomized Study.
Brief Title: Efficacy of Dicopeg Junior in Comparison With Lactulose for the Treatment of Functional Constipation in Children Aged 6 Months to 6 Years.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Medical University of Bialystok (Other); University of Rzeszow (Other)
Responsible Party: Principal Investigator, JAROSLAW KIERKUS, Ass. Prof., Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPCZD 27.01.2016
Record Dates: First submitted 2016-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Constipation
Keywords: constipation; children; polyethylene glycols (PEG); lactulose
MeSH Terms: conditions — Constipation | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dicopeg Junior (Active Comparator): Polyethylene glycols (PEG) - 3350 Dosage form: oral solution sachets Frequency: 2 doses
  Dosage:
  * weight up to 8 kg - 1 sachet per day
  * weight 8 - 12 kg - 2 sachets a day
  * weight 12 - 20 kg - 3 sachets a day
  * weight> 20 kg - 4 sachets per day, Duration: 12 weeks vs Lactulose Dosage form: oral solution Dosage: 2 ml / kg / day Frequency: 2 doses Duration: 12 weeks
  Interventions: Drug: polyethylene glycols (PEG) 3350
- Lactulose (Active Comparator): Lactulose Dosage form: oral solution Dosage: 2 ml / kg / day Frequency: 2 doses Duration: 12 weeks
  Interventions: Drug: Lactulose Oral Product

INTERVENTIONS:
Drug: polyethylene glycols (PEG) 3350 — Evaluating the efficacy of Dicopeg Junior in comparison with lactulose for the treatment of functional constipation in children aged 6 months to 6 years.
  Arms: Dicopeg Junior
Drug: Lactulose Oral Product — Evaluating the efficacy of Dicopeg Junior in comparison with lactulose for the treatment of functional constipation in children aged 6 months to 6 years.
  Arms: Lactulose

SUMMARY:
Assessment of efficacy of Dicopeg Junior, compared to lactulose, in the treatment of functional constipation in children aged 6 months to 6 years. The basis of assessment is to compare the number of commissioned stools (more than three stools per week) and stool consistency according to the scale of Bristol, in children taking Dicopeg Junior and children treated with lactulose. Childrens who meet the inclusion criteria will be randomized to one of two groups, in which the treatment will be as follows for 12 weeks:

1. The first group - Dicopeg Junior (max. in 2 doses) in a dose of:

   * weight up to 8 kg - 1 sachet per day
   * weight 8 - 12 kg - 2 sachets a day
   * weight 12 - 20 kg - 3 sachets a day
   * weight> 20 kg - 4 sachets per day,
2. The second group - Lactulose at 2 ml / kg / day (in two doses). Preparations: Dicopeg Junior and Lactulose will be administered orally for the duration of the study (12 weeks).

DETAILED DESCRIPTION:
Reason for study:

Defecation disorders, and among them constipation, are one of the most common gastrointestinal problems in children. According to data from the literature, the problem affects 1% - 7.5% of the children population who come to a general pediatrician, 25% of patients in gastroenterological practice, and even 45% in a highly specialized gastroenterology centers [1, 2]. In 17% - 40% of children with constipation symptoms begin in the first year of life [1]. The most common cause of chronic constipation in children are functional disorders, in approx. 90% of cases [3]. Essential to the diagnosis is to exclude anatomical abnormalities, neurological, endocrine and metabolic reasons, which can cause constipation, and declare at least two signs contained in the Rome III Criteria: 2 or less defecation during week, retention of large amount of fecal masses in the rectum; as well large stools which may clog the toilet [4]. The aim of treatment is to regulate bowel movements and prevent recurrence of symptoms. The mainstay of treatment is to change eating habits, defecation training and farmacotherapy with laxative drugs.

According to ESPGHAN / NASPGHAN guidelines, as first-line drugs are recommended polyethylene glycols (PEG) - 3350 or 4000, at a dose of 0.2 - 0.8 g/kg/day, and in case of unavailability or in children under 1 year of age recommends use of lactulose in a dose of 1 -3 ml/kg. Launch of preparation Dicopeg (polyethylene glycol 3350) - the first macrogol holding registration for the use of patients from 6 months of age, is giving greater therapeutic options for these patients.

In the literature, there are few reports on the use of polyethylene glycols in children. There is a need for controlled studies evaluating the efficacy and safety of use of polyethylene glycols in children, especially because that existing studies were conducted before the release of the current guidelines ESPGHAN / NASPGHAN [5].

AIM of the study:

Assessment of efficacy Dicopeg Junior for the treatment of functional constipation in children aged 6 months to 6 years.

Endpoints:

Primary Assessment of efficacy of Dicopeg Junior, compared to lactulose, in the treatment of functional constipation in children aged 6 months to 6 years. The basis of assessment is to compare the number of commissioned stools (more than three stools per week) and stool consistency according to the scale of Bristol, in children taking Dicopeg Junior and children treated with lactulose.

Secondary Assessment of the side effects of treatment, such as abdominal pain, diarrhea, nausea, vomiting, bloating, gas, irritation of the anal area. In addition, the number of stools per week, defecation with pain during the week or hard, constipated stools.

Course of study:

Day 0- inclusion in the study (first visit). Data collection which are qualifying or disqualifying the child in participation in the study and examination of the child with evaluation of fecal retention.

After examination of the patient, according to the decision of the attending physician, performing or not rectal enema cleaning prior to randomization patient.

The signing of informed consent for participation in the study by the parents of children eligible to participate in the study. Establishment a patient card (attached).

Randomization to the group with Dicopeg Junior or lactulose (central randomization).

Childrens who meet the inclusion criteria will be randomized to one of two groups, in which the treatment will be as follows for 12 weeks:

1. The first group - Dicopeg Junior (max. in 2 doses) in a dose of:

   * weight up to 8 kg - 1 sachet per day
   * weight 8 - 12 kg - 2 sachets a day
   * weight 12 - 20 kg - 3 sachets a day
   * weight> 20 kg - 4 sachets per day,
2. The second group - Lactulose at 2 ml / kg / day (in two doses). Preparations: Dicopeg Junior and Lactulose will be administered orally for the duration of the study (12 weeks).

Provide instructions concerning the use of the diary, defecation training and the use of fiber-rich diet. Issue diary, Bristol scale and test preparation.

Providing information about the possibility of telephone contact in case of diarrhea / excessive drug reaction / intolerance of the drug during the study to modify the dose.

4 weeks study Telephone consultation (on day 28 of the study) in order to monitor the status of the child, the effectiveness of treatment (number of completions stools per week, abdominal pain during defecation, stool consistency), the evaluation of side effects, discuss the entries in the diary, additional recommendations. The visit will be recorded on the patient card.

In the case of registration of intolerance or lack of efficacy of lactulose (the patient still meets the criteria Roman) in the second group it will be proposed to the patient treatment with Dicopeg Junior in accordance with the dosage in the first group to complete the 12 week study. Then the patient will be asked to come to the medical cenetr the next day, ie. in a 29 day study after receiving the preparation Lactulose.

The final 12 weeks study visit in order to evaluate the effectiveness of treatment, a summary of recommendations, assessment of adverse events and return the diary. Conducting examination. Note in the patient's diary visit.

Follow up- 16 weeks study Telephone contact to assess the state of the child, the amount of completions stools per week, abdominal pain during defecation, stool consistency, issue additional recommendations. If necessary, establish a child visits the clinic Gastrological. Note in the patient's visit.

Diary:

The table where the parent of a child writes the application preparation (Dicopeg Junior or Lactulose), the number of cast stools, their consistency, the occurrence of pain during defecation, encopresis and adverse events.

Duration:

12 weeks + 4 weeks follow-up (follow-up).

The study population. Statistics. Children aged 6 months to 6 years, fulfilling the inclusion criteria, sample size 102 patients (determined on the basis of the statistical program, taking into account the difference in the groups 30%) Assuming the difference between the groups in terms of achieving a therapeutic effect of 30%: the success of treatment group- 60% success in the control group 30%, at a power of 0.8 and assuming the test discontinuation by 20% of children final calculation of the required number of patients is 102 patients .

Assuming the difference between the groups in terms of achieving a therapeutic effect of 30%: the success of treatment group-60% success in the control group 30%, at a power of 0.8 and assuming the test discontinuation by 20% of children final calculation of the required number of patients is 102 patients .

The number of patients:

The probability of therapeutic success in the control group = 0.3 The probability of therapeutic success in test group = 0.6

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6 months - 6 years
2. Diagnosis of functional constipation according to the Rome III criteria
3. Patients newly recognized or ineffectively treated
4. Parental consent for their child's participation in the study and the way they are treatment for the duration of the study

Exclusion Criteria:

1. Well-known organic cause constipation (eg. an underactive thyroid, Hirschprung disease, cystic fibrosis).
2. Anatomical abnormality of the digestive tract.
3. Status after gastrointestinal surgery
4. Parents disagree to participate in the study
5. Intolerance of lactulose or polyethylene glycols in an interview
6. Comorbidities that may significantly affect the treatment outcome: food allergy, celiac disease, CNS disease, lactose intolerance or other disaccharide bacterial overgrowth

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy of Dicopeg Junior, compared to lactulose, in the treatment of functional constipation in children aged 6 months to 6 years. | 16 weeks
  The basis of assessment is to compare the number of commissioned stools (more than three stools per week) and stool consistency according to the scale of Bristol, in children taking Dicopeg Junior and children treated with lactulose.

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Department of Pediatrics, Gastroenterology and Allergology; Medical University of Bialystok, Bialystok
  - University of Rzeszow, Rzeszów
  - Department of Gastroenterology, Hepatology, Feeding Disorders and Pediatrics; The Childrens Memorial Health Institute, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
publication

REFERENCES:
- [Background] Tabbers MM, DiLorenzo C, Berger MY, Faure C, Langendam MW, Nurko S, Staiano A, Vandenplas Y, Benninga MA; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition; North American Society for Pediatric Gastroenterology. Evaluation and treatment of functional constipation in infants and children: evidence-based recommendations from ESPGHAN and NASPGHAN. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):258-74. doi: 10.1097/MPG.0000000000000266. PMID 24345831
- [Background] van den Berg MM, Benninga MA, Di Lorenzo C. Epidemiology of childhood constipation: a systematic review. Am J Gastroenterol. 2006 Oct;101(10):2401-9. doi: 10.1111/j.1572-0241.2006.00771.x. PMID 17032205
- [Background] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Background] Voskuijl W, de Lorijn F, Verwijs W, Hogeman P, Heijmans J, Makel W, Taminiau J, Benninga M. PEG 3350 (Transipeg) versus lactulose in the treatment of childhood functional constipation: a double blind, randomised, controlled, multicentre trial. Gut. 2004 Nov;53(11):1590-4. doi: 10.1136/gut.2004.043620. PMID 15479678
- [Derived] Jarzebicka D, Sieczkowska-Golub J, Kierkus J, Czubkowski P, Kowalczuk-Kryston M, Pelc M, Lebensztejn D, Korczowski B, Socha P, Oracz G. PEG 3350 Versus Lactulose for Treatment of Functional Constipation in Children: Randomized Study. J Pediatr Gastroenterol Nutr. 2019 Mar;68(3):318-324. doi: 10.1097/MPG.0000000000002192. PMID 30383579